CLINICAL TRIAL: NCT07021989
Title: Pembrolizumab and GVD With ctDNA-guided Consolidation in Patients With Relapsed or Refractory Classic Hodgkin Lymphoma: A Multicenter Phase 2 Study of the University of California Hematologic Malignancies Consortium
Brief Title: ctDNA-Guided Therapy for Relapsed/Refractory Hodgkin Lymphoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Michael Spinner, MD (Other)
Collaborators: UC Hematologic Malignancies Consortium (UCHMC) (Unknown); Foresight Diagnostics (Unknown); Gateway for Cancer Research (Other)
Responsible Party: Sponsor-Investigator, Michael Spinner, MD, Assistant Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25255; NCI-2025-04294 (Other: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2025-06-06; First posted 2025-06-15 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Hodgkin Lymphoma, Adult; Refractory Hodgkin Lymphoma; Classic Hodgkin Lymphoma
Keywords: circulating tumor DNA
MeSH Terms: conditions — Hodgkin Disease | interventions — pembrolizumab; Gemcitabine; Vinorelbine; liposomal doxorubicin; pegfilgrastim; Fluorodeoxyglucose F18; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Treatment (Pembrolizumab + GVD) (Experimental): All participants receive 2, 21-day cycles of 200 mg Pembrolizumab (pembro) on day 1 of each cycle (pembro) and 1000mg Gemcitabine, 20mg/m^2 of Vinorelbine, Liposomal doxorubicin 15 mg/m2 (GVD) on days 1 and 8 of each cycle for up to 2 cycles. Pegfilgrastim is administered on day 8 or 9 of each cycle. FDG-PET/CT imaging and Foresight CLARITY LDT ctDNA response after 2 cycles will determine if participants are eligible for an additional 2 cycles of pembro + GVD or salvage therapy and ASCT. Participants may be able to qualify for consolidation without ASCT (pembro and/or 30 Gy ISRT) depending on response. Radiographic response after 4 cycles will be conducted to determine eligibility for consolidation without ASCT for participants with CR or standard of care salvage therapy and ASCT, for participants with partial response (PR), stable disease (SD), or progressive disease (PD) after a second administration of pembro+GVD. Participants are followed for up to 5 years.
  Interventions: Drug: Pembrolizumab; Radiation: Non-investigational, involved site radiotherapy (ISRT); Drug: Gemcitabine; Drug: Vinorelbine; Drug: Liposomal Doxorubicin; Device: Foresight CLARITY™ LDT; Drug: Pegfilgrastim; Procedure: Fluorodeoxyglucose (FDG) Positron Emission Tomography (PET)/Computerized tomography (CT)

INTERVENTIONS:
Drug: Pembrolizumab — Given intravenously
  Other Names: Keytruda
Radiation: Non-investigational, involved site radiotherapy (ISRT) — Undergo possible, standard of care, non-investigational radiation therapy
  Other Names: ISRT
Drug: Gemcitabine — Given IV
  Other Names: Gemzar
Drug: Vinorelbine — Given IV
  Other Names: Navelbine
Drug: Liposomal Doxorubicin — Given IV
  Other Names: Doxil
Device: Foresight CLARITY™ LDT — Foresight CLARITY LDT, a laboratory-developed test (LDT),by Foresight Diagnostics, is an ultra-sensitive liquid biopsy and tissue platform that detects MRD in patients with B-cell lymphomas
  Other Names: CLARITY LDT™
Drug: Pegfilgrastim — Given IV for supportive care
  Other Names: Neulasta
Procedure: Fluorodeoxyglucose (FDG) Positron Emission Tomography (PET)/Computerized tomography (CT) — Undergo imaging
  Other Names: FDG PET/CT

SUMMARY:
This is a single arm, open-label, multicenter, phase II study of pembrolizumab (pembro), gemcitabine, vinorelbine, and liposomal doxorubicin (GVD) in patients with relapsed or refractory classic Hodgkin lymphoma (cHL) with response-adapted consolidation. This study will investigate using circulating tumor DNA (ctDNA) at pre-determined time points using Foresight CLARITY LDT, an ultra-sensitive liquid biopsy platform that detects Minimal residual disease (MRD) in patients with B-cell lymphomas using the phased variant enrichment and sequencing technology (PhasEDq) to determine response to study interventions.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the ctDNA/MRD-negative, PET-negative complete response rate for cHL patients undergoing treatment with pembro + GVD.

SECONDARY OBJECTIVES:

I. To determine progression-free survival (PFS) overall survival (OS) at 2 years among patients receiving non-transplant consolidation.

II. To determine PFS and OS at 2 years for the overall cohort.

III. To determine the proportion of patients treated with pembro + GVD and non-transplant consolidation who ultimately undergo Autologous Stem Cell Transplant (ASCT) within 2 years.

IV. To determine the rate of discordance between Positron Emission Tomography (PET)/Computerized tomography (CT) response and ctDNA/MRD response.

V. To determine the incidence of adverse events, including immune-related adverse events, in patients receiving pembro + GVD and pembrolizumab consolidation.

VI. To assess health-related quality of life (HRQOL) and patient-reported outcomes (PROs) as measured by Patient-Reported Outcomes Measurement Information System (PROMIS) 29 and Functional Assessment of Cancer Therapy-COmprehensive Score for financial Toxicity (FACIT-COST).

VII. To determine the proportion of patients with relapsed or refractory cHL for whom baseline Foresight CLARITY LDT genotyping from the peripheral blood is successful

EXPLORATORY OBJECTIVES:

I. To evaluate the kinetics of ctDNA/MRD clearance in the peripheral blood after pembro + GVD.

II. To evaluate the ctDNA/MRD-negative complete response (CR) rate and 2-year PFS stratified by cHL molecular subgroup at diagnosis (H1 vs H2 genotype).

III. To evaluate long term efficacy and toxicity outcomes for up to 5 years.

IV. To compare the performance of identification of phased variants from plasma genotyping with identification of phased variants from archival tissue genotyping.

OUTLINE:

Participants will undergo response assessment and ctDNA/MRD assessment using phased variant enrichment and detection sequencing (PhasED-Seq) using Foresight CLARITY LDT. A composite response assessment will be used to determine eligibility for non-transplant consolidation. Participants who achieve a response after 2 cycles of pembro + GVD will be eligible for non-transplant consolidation with 8 cycles of pembrolizumab and/or 30 Gray (Gy) involved-site radiotherapy (ISRT). Participants not achieving a response will discontinue study therapy and proceed to study follow-up, during which time participants can receive standard of care salvage therapy and ASCT, if eligible. Participants will be followed for up to 5 years from trial entry for long term efficacy and toxicity outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Histologically confirmed classic Hodgkin lymphoma (including nodular sclerosis, lymphocyte-rich, mixed cellularity, and lymphocyte-depleted Hodgkin lymphoma).
3. Participants must have relapsed or refractory disease after no more than one line of systemic therapy. First line therapy must have included doxorubicin.
4. At least one site of FDG-avid disease on PET/CT that is ≥ 1.5 cm in diameter for nodal disease or ≥ 1.0 cm in diameter if extranodal disease.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2 (Karnofsky ≥ 50%).
6. Demonstrates adequate organ function as defined below:

   1. Absolute neutrophil count (ANC) ≥ 1.0 X 10^9/ L (1000/microliter (mcL), growth factors permitted).
   2. Platelets ≥ 75 X 10^9 / L (75,000/mcL, platelet transfusion independent).
   3. Total bilirubin ≤ 1.5 x institutional upper limit of normal, unless elevated due to Gilbert's syndrome.
   4. Aspartate aminotransferase (AST) / (SGOT) ≤3 x institutional upper limit of normal.
   5. Alanine aminotransferase (ALT) / (SGPT) ≤3 x institutional upper limit of normal.
   6. Creatinine clearance (CrCl, calculated) ≥ 40 mL/min/1.73 m^2, calculated using the Cockcroft-Gault equation.
7. For participants with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
8. Individuals with a history of hepatitis C virus (HCV) infection must have been treated with sustained virologic response. For individuals with HCV infection who are currently on treatment, participants are eligible if there is an undetectable HCV viral load.
9. Human immunodeficiency virus (HIV)-infected individuals on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
10. Individuals with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
11. Females of reproductive potential (defined below) must be willing to undergo a urine or serum pregnancy test (i.e., human chorionic gonadotropin test) within 72 hours before start of trial therapy. A female is considered to not be of reproductive potential (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice), if the participants meet either of the following two criteria: (1) has reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause); or (2) has undergone surgical sterilization (i.e., hysterectomy and/or bilateral oophorectomy for removal of uterus and/or ovaries). The result of the urine or serum pregnancy test must be negative in order to administer initiate trial therapy. If a urine pregnancy test cannot be confirmed as negative (e.g., an ambiguous result), a serum pregnancy test is required. In such cases, the individual must be excluded from participation if the serum pregnancy result is positive. Pregnant individuals are excluded from this study because there is a potential risk for adverse effects in the unborn child secondary to treatment of the study participant with trial therapy.
12. Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

1. Participants who previously received a programmed cell death protein 1 (PD-1) inhibitor-based regimen (e.g., nivolumab or pembrolizumab + AVD) and progressed within 6 months of last done of immune checkpoint inhibitor.
2. Receipt of systemic anti-cancer therapies or radiation within 2 weeks prior to the start of trial therapy or receipt of antibody therapy within 4 weeks prior to the start of trial therapy.
3. Has participated in a study of an investigational product and received study treatment or used an investigational device within four weeks of the first dose of treatment.
4. Prior autologous or allogeneic hematopoietic stem cell transplant.
5. Systemic autoimmune disease requiring continuous immunosuppressive treatment (≥prednisone 10 mg per day or equivalent), with the exception of autoimmune thyroid disease.
6. Left ventricular ejection fraction (LVEF) <50% as assessed by transthoracic echocardiogram or multigated acquisition (MUGA) scan.
7. Participants whose lifetime cumulative dose of doxorubicin would exceed 450 mg/m^2 after receiving 4 cycles of pembro + GVD are excluded (i.e., >330 mg/m^2 at trial entry).
8. Has known hypersensitivity to pembrolizumab, gemcitabine, vinorelbine, and/or liposomal doxorubicin; or any of their excipients.
9. Has any significant medical condition or comorbidity that could compromise participants safety in the opinion of the treating investigator (e.g., uncontrolled serious infection).
10. Individuals who are pregnant or breast-feeding/chest-feeding. Pregnant and breastfeeding individuals are excluded because there is a potential risk for adverse effects in the unborn/nursing child secondary to treatment of the study participant with trial therapies. Females of reproductive potential must have a negative pregnancy test before initiation of trial therapy, as outlined in inclusion criterion #12. Breast-feeding should be discontinued before initiation of trial therapy.
11. Individuals with ongoing Grade 2 events that are not clinically stable or ongoing ≥ Grade 3 events (CTCAE v5.0 grading).
12. Notification from Foresight Diagnostics that the CLARITY LDT baseline specimen has failed sample quality control (QC) and/or the baseline ctDNA is not quantifiable. Note: Foresight will only notify sites if the specimen fails quality control (QC) or is not quantifiable. Sites will not receive notification if the specimen passes QC and is quantifiable. For QC failures, a sample re-draw may be considered upon discussion with and approval by the lead University of California, San Francisco (UCSF) Principal Investigator.
13. Individuals with any condition or social circumstance that, in the opinion of the investigator, would impair the participant's ability to comply with study activities, interfere with participant safety, or study endpoints.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-10-31 (Estimated); Primary Completion 2028-10-31 (Estimated); Study Completion 2033-04-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with a complete response | Up to 4 cycles (a cycle is 21 days)
  To determine the ctDNA/MRD negative, PET negative complete response rate for cHL, participants undergoing treatment with pembro + GVD will have a composite response incorporating the following two criteria: (1) Absence of detectable cHL ctDNA as assessed by Foresight CLARITY LDT after 2 cycles of treatment and (2) complete response by Fluorodeoxyglucose (FDG) PET/CT, assessed by Lugano criteria after 2 cycles, or 4 if participant demonstrates indeterminate response (IR) after 2 cycles. Lugano classification for response using FDG PET-CT is as follows: A score is given which ranges from 1 (No uptake above background) to 5 (Hottest area of uptake markedly > liver and/or new lesions present). A CR is defined as a score of 1,2,3 in nodal or extranodal sites with or without a residual mass. Lymphoma Response to Immunomodulatory Therapy Criteria (LYRIC) will be used to distinguish IR, SD or PD. Response rate will be summarized by percentage, along with 95% confidence intervals.

SECONDARY OUTCOMES:
Progression-free survival (PFS) rate for participants without Autologous Stem Cell Transplant (ASCT) | Up to 2 years
  PFS rate is defined as the proportion of participants alive without disease from initiation of study therapy to progression or death by any cause, whichever occurs first for up to 2 years after participants receive study therapy and non-transplant consolidation. The censoring time for PFS will be the date of the last study assessment for progression. PFS will be analyzed descriptively using Kaplan-Meier methods.
Overall Survival (OS) rate for participants without ASCT | Up to 2 years
  OS rate is defined as the proportion of participants alive from initiation of study therapy to death by any cause for up to 2 years after participants receive study therapy and non-transplant consolidation. The censoring time for OS will be the date of the last study contact. OS will be analyzed descriptively using Kaplan-Meier methods.
Overall PFS rate | Up to 2 years
  Overall PFS rate is defined as proportion of participants alive without disease from initiation of study therapy to progression or death by any cause, whichever occurs first for up to 2 years after participants receive study therapy. The censoring time for PFS will be the date of the last study assessment for progression. PFS will be analyzed descriptively using Kaplan-Meier methods.
Overall survival rate | Up to 2 years
  OS rate is defined as the proportion of participants alive from initiation of study therapy to death by any cause for up to 2 years after participants receive study therapy. The censoring time for OS will be the date of the last study contact. OS will be analyzed descriptively using Kaplan-Meier methods.
Proportion of participants undergoing ASCT | Up to 2 years
  The proportion of participants undergoing ASCT is defined as the number of participants having received an autologous stem cell graft over the total number of participants.
Percentage of participants with presence cHL ctDNA | Up to
  The percentage of participants with the presence of absence of detectable ctDNA through 2 cycles of pembro + GVD will be reported.
Percentage of participants with presence of detectable metabolically active disease | Up to 2 years
  The percentage of participants with the presence of absence of detectable metabolically active disease on an FDG PET/CT at any time during the course of treatment with Pembro+GVD will be reported.
Number of participants reporting treatment-emergent Adverse Events (AEs) of significant interest | From start of treatment until 90 days after discontinuation of treatment, approximately 2 years
  The number of participants reporting Adverse Events (AEs) will be descriptive and performed based on the safety population. Serious Adverse Events (SAEs), Immune-related Adverse Events (irAEs), AEs classified as Grade 3 or higher per NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5, and AEs resulting in discontinuation of treatment, withdrawal from the study will be tabulated.
Change in mean scores on the Patient Reported Outcomes Measurement Information System (PROMIS®-29) (Version 2) over time | Up to 5 years
  The PROMIS 29 v2.0 profile assesses pain intensity using a response scale for each item ranging from 0 (no pain) to 10 (worst imaginable pain) on seven health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance), with four items per domain and one question which addresses pain intensity item. PROMIS-29 domains are scored using a T-score metric, with higher scores indicate higher levels of functioning. Mean scores and standard deviations will be reported.
Change in mean scores on the Comprehensive Score for Financial Toxicity-Functional Assessment of Chronic Illness Therapy (COST-FACIT) survey over time | Up to 5 years
  The COST-FACIT is an 11-item measure used to assess financial toxicity. Each item is measured on a five-point Likert scale (0 = not at all, 4 = very much), with recall based on the past 7 days related to the participant's disease management. A score is computed by first reverse coding seven items, then taking the sum of all items, multiplying the sum by the number of items on the scale, and dividing that number by the number of items answered. Higher scores indicate better Financial Well-Being. Mean scores and standard deviations will be reported.
Percentage of participants with detectable cHL ctDNA at baseline | Up to 30 days
  Percentage of all participants with detectable cHL ctDNA in the plasma at baseline will be reported. Participants not meeting this criterion will be excluded from the study, but genotype failures will be recorded for the purpose of this endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Spinner, MD, Principal Investigator — University of California, San Francisco
Locations (6):
- United States (6):
  - University of California Davis, Davis, California
  - University of California San Francisco-Fresno, Fresno, California
  - University of California Irvine, Irvine, California
  - University of California, San Diego, La Jolla, California
  - Unversity of California, Los Angeles, Los Angeles, California
  - University of California, San Francisco, San Francisco, California

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared with participating research collaborators during the course of the study.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: During the course of study activities